CLINICAL TRIAL: NCT04225780
Title: The Efficiency and Safety of Low Dose IL-2 and Ganciclovir in Treatment of Cytomegalovirus Infection: an Open Label, Prospective and Control Trial
Brief Title: Treatment of Low Dose IL-2 and Ganciclovir in Cytomegalovirus Infection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLDIGCI
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Interleukin-2; Ganciclovir

STUDY DESIGN:
Intervention Model Description: We distribute the patients with CMV infection into two groups, one group will be treated with low-dose IL-2 and ganciclovir, another group will be only treated with ganciclovir.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of low-dose IL-2 and ganciclovir (Experimental): If patients are eligible, which CMV-DNA are more than 10^3 copies, it will be randomly distributed in low-dose IL-2 and ganciclovir group and low-dose IL-2 is defined as 1 million IU per day subcutaneously.
  Interventions: Drug: Low-dose IL-2 and ganciclovir
- Treatment of ganciclovir (Placebo Comparator): If patients are eligible, which CMV-DNA are more than 10^3 copies, it will be randomly distributed in ganciclovir treatment group.
  Interventions: Drug: Low-dose IL-2 and ganciclovir

INTERVENTIONS:
Drug: Low-dose IL-2 and ganciclovir — If patients are eligible, which CMV-DNA are more than 10^3 copies, it will be randomly distributed in low-dose IL-2 and ganciclovir group, or ganciclovir group. Low-dose IL-2 is defined as 1 million IU per day subcutaneously.

SUMMARY:
Cytomegalovirus (CMV) infections is a severe infection in patients of rheumatic disease treated with corticosteroid and immunosuppressive agents. Ganciclovir is the main therapy in CMV infection, accompanied with diverse side effects, including neutropenia, anemia, disorder of renal function and so on, which are also common symptoms of rheumatic diseases. Additionally, prolonged antiviral treatment may delay recovery of virus, specific immune responses, resulting in an increasing of late-onset CMV disease.

IL-2 is a pleotropic cytokine which can promote the proliferation and function of CD8+ T cells and NK cells through the combination with IL-2 receptor. Recently, several studies have revealed that low dose IL-2 is an effective and safe therapy for autoimmune disease. In systemic lupus erythematous patients, additionally, patients treated with low-dose IL-2 had lower incidence of infection with increased percentages of natural killer (NK) cells.

In this prospective clinical trial, we propose to assess the effective and safety of low-dose IL-2 combined with ganciclovir in the treatment of CMV infection. Meanwhile, we will assess the immune response of after IL-2 treatment.

DETAILED DESCRIPTION:
In rheumatic diseases, CMV infection are more frequent in patients after corticosteroid pulse treatment and long-term treatment of corticosteroid and immunosuppressor.

If patients are eligible, which CMV-DNA are more than 10^3 copies, it will be randomly distributed in low-dose IL-2 and ganciclovir group, or ganciclovir group. Low-dose IL-2 is defined as 1 million IU per day subcutaneously, The CMV-DNA levels will be monitored until it turned out to be negative. In this period, we will simultaneously monitor the immune response in regard to CMV infection, including innate immune response, such as IFN-γ, TNF-α, natural killer cells, and adaptive immune response, such as CMV specific CD8+ T cells, T helper cells and so on.

We will follow these patients for at least 3 months after drug withdrawal. If patient belonging to any of these two groups develops a viral infection, then the patient will receive treatment with ganciclovir.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Rheumatic disease by the Criteria ;
2. Patients have current CMV infection, CMV-DNA are positive.
3. Apply corticosteroid less than 1.0mg/kg/d.

Exclusion Criteria:

1. CMV-DNA is negative.
2. Other infection, such as bacteremia, hepatitis B and C viruses, HIV, syphilis, bacteremia, Epstein-Barr virus and so on.
3. Known allergies, hypersensitivity, or intolerance to IL-2 or its excipients.
4. Severe comorbidities: including 1) Heart failure (≥ grade III NYHA); 2) Renal insufficiency (creatinine clearance ≤30 ml/min); 3) Hepatic insufficiency (serum ALT or AST >3 times the ULN, or total bilirubin >ULN for the central laboratory conducting the test); 4) Other disease including hematopathy, gastrointestinal disease, endocrinopathy, pulmonary, neuropathy.
5. Malignancy.
6. Had uncontrolled psychiatric or emotional disorder.
7. Pregnant or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of NK cells cytotoxicity after treatment | Days 7 after treatment
  NK cells cytotoxicity will be detected by flow cytometry

SECONDARY OUTCOMES:
The total dose for anti-viral drugs. | Day for drug withdrawal.
  The total dose of ganciclovir
The change of cytokine after low-dose IL-2 treatment. | Day after anti-viral treatment and 3 months.
  Detect by flow cytometry and ELISA.
The change of NK cell subsets. | Day after anti-viral treatment and 3 months.
  Detect by flow cytometry.
The change of level of CMV immunoglobulin M (IgM) | Day for drug withdrawal and 3 months.
  Detect by EILSA.
The change of level of CMV immunoglobulin G (IgG) | Day for drug withdrawal and 3 months.
  Detect by EILSA.
The day for CMV infection patients convert into negative. | Days when CMV-DNA are less than 10^3 copies.
  CMV-DNA will be detected by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, PhD MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He J, Zhang R, Shao M, Zhao X, Miao M, Chen J, Liu J, Zhang X, Zhang X, Jin Y, Wang Y, Zhang S, Zhu L, Jacob A, Jia R, You X, Li X, Li C, Zhou Y, Yang Y, Ye H, Liu Y, Su Y, Shen N, Alexander J, Guo J, Ambrus J, Lin X, Yu D, Sun X, Li Z. Efficacy and safety of low-dose IL-2 in the treatment of systemic lupus erythematosus: a randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2020 Jan;79(1):141-149. doi: 10.1136/annrheumdis-2019-215396. Epub 2019 Sep 19. PMID 31537547
- See also: clinicaltrials.gov — https://www.clinicaltrials.gov/ct2/show/NCT02985775?id=NCT02505568+OR+NCT02756650+OR+NCT01960790+OR+NCT02648581+OR+NCT02985775+OR+NCT04056533+OR+NCT01185223&draw=2&rank=2&load=cart